CLINICAL TRIAL: NCT06656780
Title: Stress Inoculation Training (SIT): An Evidence-Based, Military Aligned Psychological Performance and Health Sustainment Prototype
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Department of Defense / Congressionally Mandated Research Program (CDMRP) (Unknown)
Responsible Party: Principal Investigator, Sarah Jackson, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-24-0756
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stress, Psychological
Keywords: Psychological health; resilience; Warfighter performance
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIT + Damage Control Assessment & Firefighting (DCA-FF) (Experimental)
  Interventions: Behavioral: SIT; Behavioral: DCA-FF
- DCA-FF (Active Comparator)
  Interventions: Behavioral: DCA-FF

INTERVENTIONS:
Behavioral: SIT — Participants will undergo 2 day (8 hours each) Stress Inoculation Training . This will be done in 3 steps:
  Step 1: focus on education about the human body and brain and shift to hands on skills practice to improve performance in stressful conditions and is designed to improve self-and-situational awareness and the ability to manipulate reactions and responses in the body on purpose to enhance performance
  Step 2: focuses on improving mental self-awareness and gaining skills in Mental Agility and Mental Flexibility
  Step 3: participants will have specific simulations and real-world opportunities to practice the skills learnt.
  Arms: SIT + Damage Control Assessment & Firefighting (DCA-FF)
Behavioral: DCA-FF — Participants will undergo 8-week Standard Firefighting Training

SUMMARY:
The purpose of this study is to demonstrate the feasibility of augmenting existing/traditional Navy military training with the manualized SIT Core Protocol (CP) utilizing the established augmentation procedure set as measured by feasibility, utility, and satisfaction metrics (CSQ-8) and to examine the relative effectiveness of the SIT-CP by comparison to standard military training in a controlled trial examining outcomes of stress tolerance, psychological health, resilience and occupational performance in Sailors undergoing DCA Firefighting Training (pre- to post-training), while collecting implementation data.

ELIGIBILITY:
Inclusion Criteria:

* US Navy service members on Active Duty or Reserve status
* be fluent in English.
* be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
* have access to a SmartPhone, computer, or tablet to utilize and access the virtual classroom.
* agree to undergo psychometric and operational performance testing and participate in ongoing assessments throughout the study duration.
* be willing to comply with all study procedures, able to complete all assessments independently, and available for the duration of the study (with reasonable accommodations for military operational demands as they arise).

Exclusion Criteria:

* Active suicidal ideation as assessed by the Investigator at screening or as identified during the study.
* Clinically significant history of psychotic disorder, bipolar spectrum disorder, or neurodegenerative disease/dementia as assessed by the Investigator.
* Active severe substance abuse as assessed by the investigator in accordance with The Diagnostic and Statistical Manual of Mental Illnesses (DSM-5) Substance Abuse Disorder criteria, or presence of illicit substance abuse.
* They are currently undergoing another form of treatment other than supportive therapy (>2 times per month).
* Any other condition/situation that the Investigator believes may interfere with participant safety, study conduct, or interpretation of study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in perceived management of stress as assessed by the Perceived Stress Scale (PSS) | Baseline, about 3 weeks from baseline, about 6 weeks form baseline, about 11 weeks form baseline, end of study (an average of 19 weeks form baseline)
  This is a 10 item questionnaire and each is scored a 5 -point likert scale from 0(never) to 4(very often) for a score range of 0 to 40, higher total scores indicate higher perceived stress.
Change in resilience as assessed by the Connor-Davidson Resilience Scale (CD-RISC) | Baseline, about 3 weeks from baseline, about 6 weeks form baseline, about 11 weeks form baseline, end of study (an average of 19 weeks form baseline)
  This is a 25 item questionnaire and each is scored on a 5-point Likert scale ranging from 0 (Not true at all) to 4 (True nearly all the time) for a maximum score of 100 higher score indicating more resilience

SECONDARY OUTCOMES:
Successful presentation of the element in the training module as assessed by the SIT Feasibility Rubric | week 2
  This is a is a dichotomous measure (1-successful vs. 0-unsuccessful)
Successful presentation of the element in the training module as assessed by the SIT Feasibility Rubric | week 4
  This is a is a dichotomous measure (1-successful vs. 0-unsuccessful)
level of confidence with delivering the training elements within the Module and the full Module as assessed by the SIT Feasibility Rubric | week 2
  This is scored on a likert scale from 1(low) to 5(high)
level of confidence with delivering the training elements within the Module and the full Module as assessed by the SIT Feasibility Rubric | week 4
  This is scored on a likert scale from 1(low) to 5(high)
Utility as assessed by the standardized self-assessment tool | week 2
  high utility is when greater than 80% of novice SIT Trainers reporting an average of >80% on standardized self-assessment rubrics of protocol Module delivery.
Utility as assessed by the standardized self-assessment tool | week 4
  high utility is when greater than 80% of novice SIT Trainers reporting an average of >80% on standardized self-assessment rubrics of protocol Module delivery.
Satisfaction as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8) | week 2
  This is an 8 item questionnaire and each is scored on a 4-point Likert scale ranging from 1 (lowest satisfaction) to 4 (highest satisfaction) for a score range of 8 to 32, higher score indicating more satisfaction
Satisfaction as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8) | week 3
  This is an 8 item questionnaire and each is scored on a 4-point Likert scale ranging from 1 (lowest satisfaction) to 4 (highest satisfaction) for a score range of 8 to 32, higher score indicating more satisfaction
Satisfaction as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8) | week 11(end of study)
  This is an 8 item questionnaire and each is scored on a 4-point Likert scale ranging from 1 (lowest satisfaction) to 4 (highest satisfaction) for a score range of 8 to 32, higher score indicating more satisfaction
Firefighting Observational Rubrics | week 6
  These are observational rubrics, utilized by the firefighting instructors to evaluate occupational performance of the participants on specific firefighting task
Change in adaptation to stress as assessed by the Situational Adaptation to Stress Scale for Human Performance (SASS-HP) | Baseline, about 3 weeks from baseline, about 6 weeks form baseline
  The premeasurement scale is a 9 item questionnaire and each is scored on a likert scale from 1(totally disagree) -5(totally agree), higher score indicates better outcome
Change in adaptation to stress as assessed by the Situational Adaptation to Stress Scale for Human Performance (SASS-HP) | about 11 weeks form baseline, end of study (about 19 weeks form baseline)
  The post measurement scale is a 18 item questionnaire and each is scored on a likert scale from 1(totally disagree) -5(totally agree), higher score indicates better outcome
Change in mental skills as assessed by the Test of Performance Strategies (TOPS) | Baseline, about 6 weeks form baseline, about week 11, end of study (19 weeks form baseline)
  This is a 68 item questionnaire and each is scored on a 5-point Likert scale from 1(never) to 5(always) for a maximum score of 340 , higher score indicating better outcome
Change in achievement score as assessed by the 10-Minute Heart Rate Variability Biofeedback assessment Assessment | Baseline, week 11
  Achievement score is based on an algorithm that uses variability in heart rate over time and heart beats per minute. It indicates percentage of time participant is able to relax.The score range is 0-500+. Higher score means better outcome
Change in average coherence as assessed by the 10-Minute Heart Rate Variability Biofeedback assessment Assessment | Baseline, week 11
  Coherence score is based on an algorithm that uses variability in heart rate over time and heart beats per minute. It indicates percentage of time participant is able to relax.The score range is 0-500+. Higher score means better outcome
Change in average heart beats per minute as assessed by the 10-Minute Heart Rate Variability Biofeedback assessment | Baseline, week 11
  Lower heart beats is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jackson, MFT, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No